CLINICAL TRIAL: NCT01068145
Title: Randomized, Double-Blind, Multiple-Dose, Placebo-Controlled, Incomplete Crossover, Two-Part Study to Evaluate the Dose Response of SCH 527123 on Sputum Neutrophilia Following Ozone Challenge in Healthy Subjects and COPD Patients
Brief Title: Two-Part Study to Evaluate the Dose Response of SCH 527123 on Sputum Neutrophilia Following Ozone Challenge in Healthy Subjects and Chronic Obstructive Pulmonary Disease (COPD) Patients (P05567 AM7)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: P05567; 2008-006650-18 (EudraCT Number)
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 2-hydroxy-N,N-dimethyl-3-(2-((1-(5-methylfuran-2-yl)propyl)amino)-3,4-dioxocyclobut-1-enylamino)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Very low dose SCH 527123 (Experimental)
  Interventions: Drug: SCH 527123
- Low dose SCH 527123 (Experimental)
  Interventions: Drug: SCH 527123
- Medium dose SCH 527123 (Experimental)
  Interventions: Drug: SCH 527123
- High dose SCH 527123 (Experimental)
  Interventions: Drug: SCH 527123
- Placebo to match SCH 527123 (Placebo Comparator)
  Interventions: Drug: Placebo
- Low dose SCH 527123 (Part 2) (Experimental)
  Interventions: Drug: SCH 527123
- Medium dose SCH 527123 (Part 2) (Experimental)
  Interventions: Drug: SCH 527123
- High dose SCH 527123 (Part 2) (Experimental)
  Interventions: Drug: SCH 527123
- Placebo (Part 2) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCH 527123 — Very low dose SCH 527123, once daily for 7 days
  Arms: Very low dose SCH 527123
Drug: SCH 527123 — Low dose SCH 527123, once daily for 7 days
  Arms: Low dose SCH 527123
Drug: SCH 527123 — Medium dose SCH 527123, once daily for 7 days
  Arms: Medium dose SCH 527123
Drug: SCH 527123 — High dose SCH 527123, once daily for 7 days
  Arms: High dose SCH 527123
Drug: Placebo — Placebo capsules to match SCH 527123, once daily for 7 days
  Arms: Placebo to match SCH 527123
Drug: SCH 527123 — Low dose capsule SCH 527123, once daily for 14 days
  Arms: Low dose SCH 527123 (Part 2)
Drug: SCH 527123 — Medium dose capsule SCH 527123, once daily for 14 days
  Arms: Medium dose SCH 527123 (Part 2)
Drug: SCH 527123 — High dose capsule SCH 527123, once daily for 14 days
  Arms: High dose SCH 527123 (Part 2)
Drug: Placebo — Placebo capsules to match SCH 527123, once daily for 14 days
  Arms: Placebo (Part 2)

SUMMARY:
Trial to evaluate the dose response of SCH 527123 in reducing inflammation from an ozone-induced sputum neutrophilia in both healthy subjects and subjects with COPD.

ELIGIBILITY:
Inclusion Criteria:

Part 1

* Subject of either sex and of any race between the age of 18 and 55 years, with a BMI (weight [kg]/height [m2]) between 19 and 32.
* Subject must have a FEV1 ≥ 80 % of predicted value.
* Subject must be nonsmoker (including cigarettes, cigars and pipes) or exsmoker who has stopped smoking for at least 6 months (smoking history ≤ 5 pack years).
* Subject's clinical laboratory tests (CBC, blood chemistry, urinalysis) must be within normal limits. Subjects must have a neutrophil count of >2.0 x 109/L. (also Part 2)
* Subject must be free of any clinically significant disease that would interfere with the study evaluations (also Part 2).
* Screening ECG conduction intervals must be within gender specific normal range; QTcB males ≤430 msec and females ≤450 msec (also Part 2).
* Vital sign measurements must be: a) oral body temperature, between 35.0°C and 37.5°C; b) systolic blood pressure, 90 to 140 mm Hg (160 mm Hg, Part 2); c) diastolic blood pressure, 45 to 90 mm Hg (100 mm Hg, Part 2); d) pulse rate, 40 to 100 bpm.
* Subject and partner(s) must be using an accepted method of contraception during the trial through 2 months post-treatment (also Part 2).
* Prior to randomization, subject must be a responder to ozone (also Part 2).

Part 2

* Subject with a diagnosis of COPD for at least 1 year and FEV1 ≥65% of predicted value post bronchodilation (measurement 30 minutes after 400 mcg salbutamol administration) and FEV1/FVC of <70%.
* Subject of either sex and of any race between the age of 40 and 65 years, with a BMI between 19 and 32.
* Subject must be active or exsmoker (cigarettes, cigars and/or pipes).
* Subject must have a normal exercise stress test (no clinically significant ECG findings).

Exclusion Criteria:

Part 1 and Part 2

* Female subject who is pregnant, intends to become pregnant (within 3 months of ending the study), or is breastfeeding.
* Subject with history of seasonal or perennial allergic rhinitis (ie, season for specific allergen).
* Subject who has an allergy or a contraindication to excipients in placebo or SCH 527123 formulations or salbutamol.
* Surgical or medical condition (history or presence) which might alter the ADME of the drug: a) inflammatory bowel disease, ulcers, gastrointestinal or rectal bleeding; b) major gastrointestinal tract surgery, ie, gastrectomy, gastroenterostomy, or bowel resection; c) pancreatic injury or pancreatitis; d) liver disease or injury; e) impaired renal function indicated by abnormal creatinine, urinary albumin, BUN/urea or clinical significant urinary cellular constituents (eg, cast); or f) urinary obstruction or difficulty in voiding.
* Subject who has any infectious disease within 4 weeks prior to drug administration.
* Subject who is positive for hepatitis B surface antigen, hepatitis C antibodies or HIV.
* Subject who has a positive screen for drugs with a high potential for abuse (Screening and/or treatment period).
* Subjects with a history of mental instability or who have been treated for mood disorder.
* Subject with a history of alcohol or drug abuse in the past 2 years.
* Subject who has donated blood in the past 60 days.
* Subject who has demonstrated allergic reactions (eg, food, drug, atopic reactions or asthmatic episodes) which may interfere with ability to participate in the trial.
* Subject who has previously received SCH 527123 (Part 2 only)
* Subject who has received any of the following treatments more recently than indicated washout period prior to Baseline:

  * Parts 1 and 2: OTC medications (excluding paracetamol), 14 days.
  * Part 1: prescription medications, 14 days; investigational drugs, 30 days.
  * Part 2: vitamins and herbal supplements, 14 days; statins, 4 weeks; steroids (inhaled), 4 weeks; steroids (oral and dermal), 8 weeks; antibiotics, 6 weeks; leukotriene antagonists, 4 weeks; NSAIDS, 2 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
PD/PK: Dose response of SCH 527123 on ozone-induced sputum neutrophilia in healthy subjects (Part 1) and subjects with COPD (Part 2), measured by placebo-adjusted percent change in sputum neutrophil counts and absolute sputum neutrophil counts. | Part 1, four treatment periods, Part 2 three treatment periods duration of the trial.

REFERENCES:
- [Result] Holz O, Khalilieh S, Ludwig-Sengpiel A, Watz H, Stryszak P, Soni P, Tsai M, Sadeh J, Magnussen H. SCH527123, a novel CXCR2 antagonist, inhibits ozone-induced neutrophilia in healthy subjects. Eur Respir J. 2010 Mar;35(3):564-70. doi: 10.1183/09031936.00048509. Epub 2009 Jul 30. PMID 19643947